CLINICAL TRIAL: NCT00001050
Title: Women's AIDS Cohort Study (WACS)
Brief Title: Study of Women Who Have AIDS
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: WACS
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To study the effect of pregnancy, age, drug use, and coinfections on HIV progression rate. To document the prevalence, incidence, characteristics, and course of HIV infection and anogenital intraepithelial neoplasia among HIV-positive and HIV-negative women. To study the effect of HIV disease on gynecologic health including infections and reproductive function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY - Brooklyn, Brooklyn, New York, United States

REFERENCES:
- [Background] Bassuk SS, Albert CM, Cook NR, Zaharris E, MacFadyen JG, Danielson E, Van Denburgh M, Buring JE, Manson JE. The Women's Antioxidant Cardiovascular Study: design and baseline characteristics of participants. J Womens Health (Larchmt). 2004 Jan-Feb;13(1):99-117. doi: 10.1089/154099904322836519. PMID 15006283
- [Background] Mason PJ, Manson JE, Sesso HD, Albert CM, Chown MJ, Cook NR, Greenland P, Ridker PM, Glynn RJ. Blood pressure and risk of secondary cardiovascular events in women: the Women's Antioxidant Cardiovascular Study (WACS). Circulation. 2004 Apr 6;109(13):1623-9. doi: 10.1161/01.CIR.0000124488.06377.77. Epub 2004 Mar 15. PMID 15023883